CLINICAL TRIAL: NCT05680688
Title: Conditioned Pain Modulation Effects of Manual Therapy in University Students With Recurrent or Chronic Neck Pain
Brief Title: Effects of Painful Compared to Painless Manual Therapy on Pain Processing in University Students With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josue Fernandez Carnero (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PAINMT1
Record Dates: First submitted 2022-12-27; First posted 2023-01-11 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Neck Pain
Keywords: Manual Therapy; Physiotherapy; Physical Therapy; Conditioned Pain Modulation; Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Painful Manual Therapy (Experimental): Manual therapy treatment shall be carried out at a high intensity that causes pain to the patient. The aim is to provoke a medium intensity pain to the patient of 5/10 in the NRS. The physiotherapist will ask every 30 seconds the pain provoked by the treatment with the numeric rating scale (NRS) and the patient will give continuous feedback. Based on this, the physiotherapist will adapt the intensity of the treatment to provoke a medium intensity pain.
  Interventions: Other: Manual Therapy
- Painless Manual Therapy (Active Comparator): Manual therapy treatment shall be performed at a low intensity that does not cause pain to the patient. The aim is for the patient to report a pain intensity of 0/10 in NRS throughout treatment. The physiotherapist will ask every 30 seconds the pain provoked by the treatment with NRS and the patient will give continuous feedback. Based on this, the physiotherapist will adapt the intensity of the treatment to be performed below the pain threshold.
  Interventions: Other: Manual Therapy

INTERVENTIONS:
Other: Manual Therapy — * Postero-anterior mobilizations: the physiotherapist will place his thumbs on the posterior surface of the spinous process of the vertebra previously assessed as the most painful to mobilise. The oscillations will be performed at the frequency of 1 oscillation per second and will be performed 3 series of 3 minutes, with a 1 minute rest interval.
  * Pressure: The point of greatest pain shall be treated by maintained pressure in each of the following areas: right upper trapezius, left upper trapezius, right paravertebral musculature and left paravertebral musculature. Pressure shall be applied to each of the points for 1 minute.
  * Massage: Pressure is applied to the muscles by sliding along the muscle belly. This will be done slowly to control the pain that is being provoked. 3 minutes will be carried out on each upper trapezius, sliding from the acromion to the occipital and another 3 minutes on the paravertebral musculature on each side, sliding from T1 to the occipital.

SUMMARY:
The purpose of this study is to evaluate the effects of provoking pain with manual therapy on pain processing in university students with recurrent or chronic neck pain.

DETAILED DESCRIPTION:
The mechanical stimulus produced in manual therapy (MT) techniques elicits neurophysiological responses within the peripheral and central nervous system responsible for pain inhibition. Almost all types of MT elicit a neurophysiological response that is associated with the descending pain modulation circuit. But it has not been demonstrated whether this inhibition occurs through a conditioned pain modulation mechanism generated by the pain that manual therapy techniques may elicit in the patient.

ELIGIBILITY:
Inclusion Criteria:

* University students
* Chronic neck pain (persistent pain > 3 months almost every day of the week) or recurrent neck pain (repeated episodes of neck pain starting > 3 months ago with pain-free periods)
* Non-specific neck pain (pain in the neck region that is not attributable to a known specific such as herniated disc, myelopathy, fractures, spinal stenosis, neoplasm etc. nor is it associated with traumatic causes such as whiplash)
* Mean NRS score the last week > 2/10 and presence of pain on the day of assesment and treatment

Exclusion Criteria:

* Signs of radiculopathy or neuropathic pain
* Neck surgeries
* Inflammatory rheumatic
* Neurological, cardiorespiratory, oncological or psychiatric disease
* Pregnancy
* Not being able to read Spanish in order to fill in the questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Tibialis Anterior Pressure Pain Threshold (PPT) to immediate post-intervention | At baseline and immediately after the intervention
  PPTs will be assessed bilaterally (the mean between both sides will be used for analysis) over the tibialis anterior muscle (remote pain-free area) using a digital algometer (Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials for each side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.
Change from Baseline in extensor carpi ulnaris PPT to immediate post-intervention | At baseline and immediately after the intervention
  PPTs will be assessed bilaterally (the mean between both sides will be used for analysis) over the extensor carpi ulnaris muscle (remote pain-free area) using a digital algometer (Model FPX, Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials for each side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.
Change from Baseline in upper trapezius PPT to immediate post-intervention | At baseline and immediately after the intervention
  PPTs will be assessed bilaterally (the mean between both sides will be used for analysis) over the extensor upper trapezius muscle (symptomatic area) using a digital algometer (Model FPX, Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials for each side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.
Change from Baseline in spinous process of C7 PPT to immediate post-intervention | At baseline and immediately after the intervention
  PPT will be assessed over the spinous process of C7 (cervical innervated-related area) using a digital algometer (Model FPX, Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.

SECONDARY OUTCOMES:
Change from Baseline in Pain Intensity by Numeric Rating Scale (NRS) to immediate post-intervention | At baseline and immediately after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 4 hours post-intervention | At baseline and 4 hours after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 1 day post-intervention | At baseline and 1 day after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 2 days post-intervention | At baseline and 2 days after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 3 days post-intervention | At baseline and 3 days after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 4 days post-intervention | At baseline and 4 days after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 5 days post-intervention | At baseline and 5 days after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 6 days post-intervention | At baseline and 6 days after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Change from Baseline in Pain Intensity by NRS to 7 days post-intervention | At baseline and 7 days after the intervention
  The NRS measures the pain intensity using a 11-point scale. Rank from 0 to 10, with the 0-end point labeled with "no pain" and the 10-end point labeled as "worst imaginable pain".
Self-perceived improvement by Global Rating of Change (GROC scale) immediately after the intervention | Immediately after the intervention
  The GROC assesses self-perceived improvement on a scale from -7 (a very great deal worse) to +7 (a very great deal better).
Self-perceived improvement by Global Rating of Change (GROC scale) 7 days after the intervention | 7 days after the intervention
  The GROC assesses self-perceived improvement on a scale from -7 (a very great deal worse) to +7 (a very great deal better).
Change from Baseline in Parallel Conditioned Pain Modulation (CPM) to immediate post-intervention | At baseline and immediately after the intervention
  To evaluate conditioned pain modulation (CPM), a handheld pressure algometer will be used as the test stimulus to evaluate the PPT at the nail bed of the thumb of the symptomatic side before and during application of a conditioning stimulus. Ischemic muscle pain will be used as the conditioning stimulus using a sphygmomanometer. The sphygmomanometer will be applied around the upper arm of the asymptomatic side, with its lower rim 3 cm proximal to the cubital fossa. The cuff was inflated to 260 mmHg and maintained until the subject perceived a 7/10 pain on the NRS. The CPM will be the result of the PPT during the conditioning stimulus minus the PPT before the conditioning stimulus.
Change from Baseline in Sequential Conditioned Pain Modulation (CPM) to immediate post-intervention | At baseline and immediately after the intervention
  To evaluate conditioned pain modulation (CPM), a handheld pressure algometer (Model FPX, Wagner instruments, Greenwich, CT, USA) will be used as the test stimulus to evaluate the PPT at the nail bed of the thumb of the symptomatic side before and 1 minute after application of a conditioning stimulus. Ischemic muscle pain will be used as the conditioning stimulus using a sphygmomanometer. The sphygmomanometer will be applied around the upper arm of the asymptomatic side, with its lower rim 3 cm proximal to the cubital fossa. The cuff was inflated to 260 mmHg and maintained until the subject perceived a 7/10 pain on the NRS. The CPM will be the result of the PPT after the conditioning stimulus minus the PPT before the conditioning stimulus.
Change from Baseline in Termporal Summation of Pain (TSP) to immediate post-intervention | At baseline and immediately after the intervention
  TSP will be elicited with 10 applications of the algometer (Model FPX, Wagner instruments, Greenwich, CT, USA) at the individual PPT intensity perceived at the nail bed of the thumb of the asymptomatic side. For each pulse, the pressure will be increased at a rate of approximately 2 kg/second to the previously determined PPT intensity. Pulses will be presented with an interstimulus interval of 1 second because this has previously been shown to be optimal for inducing TSP with pressure pain. Before application of the first pressure pulse, subjects were instructed to manually rate the pain intensity of the first and 10th pulse with a NRS. The TSP will be calculated as the difference between the pain intensity of the tenth stimulus minus the first stimulus.
Change from Baseline in Cold Pain Intensity to immediate post-intervention | At baseline and immediately after the intervention
  Cold pain intensity will be evaluated with the subject resting on a chair with the ice application test. Testing will be conducted on the anterior skin of the right forearm.
  For the ice application test, the ice pack will be held on the skin for 10 s. After 10 s of ice application, subjects will be instructed to rate the intensity of pain on NRS. The procedure will be repeated three times to obtain a mean value, with a 60 s rest period between measures to avoid summation of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bialosky JE, Beneciuk JM, Bishop MD, Coronado RA, Penza CW, Simon CB, George SZ. Unraveling the Mechanisms of Manual Therapy: Modeling an Approach. J Orthop Sports Phys Ther. 2018 Jan;48(1):8-18. doi: 10.2519/jospt.2018.7476. Epub 2017 Oct 15. PMID 29034802
- [Background] Vigotsky AD, Bruhns RP. The Role of Descending Modulation in Manual Therapy and Its Analgesic Implications: A Narrative Review. Pain Res Treat. 2015;2015:292805. doi: 10.1155/2015/292805. Epub 2015 Dec 16. PMID 26788367
- [Background] Melzack R. Prolonged relief of pain by brief, intense transcutaneous somatic stimulation. Pain. 1975 Dec;1(4):357-373. doi: 10.1016/0304-3959(75)90073-1. PMID 141644
- [Background] WAND-TETLEY JI. Historical methods of counter-irritation. Ann Phys Med. 1956 Jul;3(3):90-9. doi: 10.1093/rheumatology/iii.3.90. No abstract available. PMID 13363246